CLINICAL TRIAL: NCT04692493
Title: A Real-World Comparative Effectiveness Trial of Treatment Strategies in Patients With Rheumatoid Arthritis: The RA-PRO Pragmatic Trial (RA-PROPR)
Brief Title: RA-PRO PRAGMATIC TRIAL
Acronym: RA-PROPR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jasvinder A Singh, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300006596; CER-2020C1-19193 (Other Grant/Funding Number: PATIENT-CENTERED OUTCOMES RESEARCH INSTITUTE (PCORI))
Record Dates: First submitted 2020-12-15; First posted 2020-12-31 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- targeted synthetic DMARD class (Active Comparator): Switching to a targeted synthetic DMARD (choice from targeted synthetic DMARDs; currently available are tofacitinib, baricitinib, upadacitinib) in people with active RA despite current treatment
  Interventions: Drug: targeted synthetic DMARD class
- non-TNFi-biologic class (Active Comparator): Switching to a non-TNFi-biologic (choice from non-TNFi-biologics; currently available are rituximab, abatacept, tocilizumab, or sarilumab) in people with active RA despite current treatment,
  Interventions: Drug: non-TNFi-biologic class

INTERVENTIONS:
Drug: targeted synthetic DMARD class — Switching to a targeted synthetic DMARD (choice from targeted synthetic DMARDs; currently available are tofacitinib, baricitinib, upadacitinib) in people with active RA despite current treatment
  Arms: targeted synthetic DMARD class
Drug: non-TNFi-biologic class — Switching to a non-TNFi-biologic (choice from non-TNFi-biologics; currently available are rituximab, abatacept, tocilizumab, or sarilumab) in people with active RA despite current treatment,
  Arms: non-TNFi-biologic class

SUMMARY:
The 2021 ACR RA treatment guideline, based on widely acknowledged low to moderate quality evidence, recommends switching to a non-tumor necrosis factor (TNFi) biologic (choose among existing medications, currently, rituximab, abatacept, tocilizumab, or sarilumab) or a targeted synthetic DMARD arm (tsDMARD; choose among existing medications, currently, tofacitinib, baricitinib, upadacitinib) in patients with active RA despite the use of a TNFi-biologic. In practice, most patients receive another TNFi-biologic, i.e., a second TNFi-biologic first. This is not based on solid evidence, but on arbitrary algorithms often proposed by health insurance plans, and/or physician experience and habit (TNFis launched 22 yrs ago vs. the first tsDMARD 8 years ago vs. first non-TNF-biologic launched 17 years ago). This study will fill a critical knowledge gap by generating CER data for important PROs between these treatment options, switching to a non-TNFi biologic or a tsDMARD in patients with active RA despite the use of a TNFi-biologic.

DETAILED DESCRIPTION:
Treatment of RA with a non-TNFi biologic (rituximab, abatacept, tocilizumab, or sarilumab) was associated with improved function, quality of life, and productivity. TsDMARDs (tofacitinib, baricitinib, upadacitinib) were similarly effective. No meaningful differences were noted in non-TNFi-biologic vs. tsDMARD, but head-to-head studies of biologics are lacking. HAQ is a sensitive outcome for RA trials. A PCORI systematic review for early RA treatment concluded that "Evidence was insufficient to evaluate any differences between biologics for their impact on either functional capacity or HRQOL", a key knowledge gap our study will fill.

The 2021 ACR RA treatment guideline, based on widely acknowledged low to moderate quality evidence, recommends switching to a non-TNFi biologic or a tsDMARD in patients with active RA despite the use of a TNFi-biologic. In practice, most patients receive another TNFi-biologic first, i.e., a second TNFi. This is not based on solid evidence, but on arbitrary algorithms often proposed by health insurance plans, and physician experience (first TNFi launched 22 yrs ago vs. the first tsDMARD 8 yrs ago vs. first non-TNF-biologic launched 17 years ago). This study will fill a critical knowledge gap by generating CER data for important PROs between these treatment options. This will facilitate informed decision-making, since PROs may be more sensitive to different mechanisms of action, and are highly relevant to patients.

The proposed study will also provide needed evidence for real-world treatment decisions made by public and private payers. This head-to-head pragmatic trial will be the first to provide CER data for improvement in key PROs with recommended strategies in active RA despite the use of a TNFi-biologic and addresses PCORI and IOM priority areas by comparing the two most commonly used RA treatment strategies for people with active RA despite the use of a TNFi-biologic. This research is patient-centered, as study outcomes were identified by patients and payers. Currently, treatment choices are based on physician experience and insurance payer limitations. Investigators will generate evidence to help patients make decisions for themselves based on outcomes they care most about based on the relative efficacy of outcomes.

Investigators will: (1) compare improvements in PROs with RA treatment strategies to each other using a state-of-the-art real-world pragmatic effectiveness study design, which will for the first time include most RA patients with comorbidities;(2) compare their toxicity in a real-world population for TNFi-biologic vs. tsDMARD. To our knowledge, no previous RCT comparing these drugs has examined a PRO as a primary outcome in RA, which our study will pioneer by using HAQ. HAQ is sensitive to change with effective treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with active, disabling RA (CDAI ≥10 and HAQ ≥0.5) despite the use/experience of a TNFi-biologic OR discontinued the medication(s) due to intolerability or toxicity irrespective of treatment duration prior to the first dose of study drug ;
2. If receiving glucocorticoids (≤10 mg/day of prednisone of equivalent) or NSAIDs, on stable doses for ≥2 weeks prior to randomization; and
3. Insurance plan or patient assistance program allows access to at least 1 drug in each of the two treatment strategies, TNFi-biologic vs. tsDMARD.(TNFi-biologic and tsDMARD) will be obtained through insurance plan or a patient assistance program/plan.

Participants will be allowed to continue their conventional synthetic DMARD (csDMARD) therapy if they had been using it for ≥ 3 months and on a stable dose for ≥ 4 weeks prior to the first dose of study drug. The following csDMARDs are allowed: methotrexate (MTX), sulfasalazine, hydroxychloroquine, and leflunomide

Exclusion Criteria:

1. Prior treatment with more than three biologics, defined as TNFi-biologic or non-TNFi biologic
2. Prior treatment with targeted synthetic DMARD
3. Concomitant use of leflunomide, sulfasalazine, cyclosporine, or azathioprine within 2-months before randomization;
4. History of sensitivity to all 4 non-TNF-biologic or a targeted synthetic DMARD;
5. Glucocorticoid injection (intravenous, intramuscular, or intraarticular) within 1 month of study entry;
6. Live vaccine within 90 days of study entry;
7. Acute or chronic infections with parenteral antibiotics or hospitalization (including tuberculosis, bacterial sepsis; invasive fungal infections (such as histoplasmosis)) within 1 month or oral antibiotics within 2 weeks of study entry;
8. History of HIV or any opportunistic infection;
9. New York Heart Association Class III or IV heart failure;
10. Latent TB for which anti-tubercular treatment has not been started;
11. Untreated Hepatitis B or C infection;
12. History of deep venous thrombosis or pulmonary embolism; or
13. Pregnant or nursing women; or
14. History of herpes zoster or shingles in the previous 12 months and not subsequently vaccinated with herpes zoster vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 924 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Limitation | Change from baseline to 12 months
  Function limitation assessed by Health assessment questionnaire (HAQ); HAQ assesses difficulty in 20 items in 8 categories (dressing, arising, eating, walking, hygiene, reaching, gripping, and outside activity), the total score ranges from 0 (no disability) to 3 (complete disability). Higher score is worse, and indicates poor function.

CONTACTS AND LOCATIONS:
Overall Officials: Jasvinder Singh, MD, Principal Investigator — University of Alabama at Birmingham
Locations (49):
- United States (48):
  - East Alabama Arthritis Center PC, Auburn, Alabama
  - Bendcare, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - SunValley Arthritis Center, Ltd, Peoria, Arizona
  - University of Arizona, Tucson, Arizona
  - Pacific Arthritis Care Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Arthritis Medical Center, Nipomo, California
  - Turlock Arthritis & Osteoporosis Center,, Turlock, California
  - Center for Rheumatology Research, Woodland Hills, California
  - George Munoz MD, PC, Aventura, Florida
  - American Arthritis and Rheumatology Associates LLC, Clearwater, Florida
  - CZ Rheumatology, Coral Springs, Florida
  - American Arthritis and Rheumatology Associates LLC, Fort Lauderdale, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Palm Beach Rheumatology and Wellness, Jupiter, Florida
  - Arthritis & Rheumatology Center of South Florida, Margate, Florida
  - Life Medical Research Group, Miami Gardens, Florida
  - Southwest Florida Rheumatology, Riverview, Florida
  - Southeast Georgia Physician Associates-Rheumatology, Brunswick, Georgia
  - Indiana University Health, Carmel, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts University, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - American Arthritis and Rheumatology Associates -Mi PLLC, Okemos, Michigan
  - Saint Paul Rheumatology, P.A., Eagan, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Dr. Jayashree Sinha, Clovis, New Mexico
  - Inspire Santa Fe Medical Group, Santa Fe, New Mexico
  - New York University, New York, New York
  - Hospital for Special Surgery, New York, New York
  - University Hospital Cleveland Medical Ctr, Cleveland, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - Arthritis and Rheumatology of Southwest Ohio, Liberty Township, Ohio
  - Southern Ohio Rheumatology, Wheelersburg, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Rheumatology and Arthritis Care Center, Exton, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - PA Regional Center for Arthritis and Osteoporosis Research, Wyomissing, Pennsylvania
  - Cumberland Rhematology, Crossville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Heritage Rheumatology and Arthritis Care, Colleyville, Texas
  - Southwest Medical Center, Dallas, Texas
  - Texas Arthritis Center, PA, El Paso, Texas
  - American Arthritis and Rheumatology Associates-Tx PLLC, Harlingen, Texas
  - Baylor University, Houston, Texas
  - Northern Virginia Center for Arthritis-Reston, Reston, Virginia
- Mount Sinai Hospital (Canada), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No